CLINICAL TRIAL: NCT05937815
Title: Monitoring of the Intestine-lung Axis of Cystic Fibrosis Patients Treated With the Combination Elexacaftor/Tezacaftor/Ivacaftor: Study of the Pulmonary and Gut Microbiota and Inflammation
Brief Title: Intestine-lung Axis of Cystic Fibrosis Patients Treated With the Combination Elexacaftor/Tezacaftor/Ivacaftor
Acronym: KAF-BIOTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2021/14
Record Dates: First submitted 2023-06-27; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis
Keywords: elexacaftor/tezacaftor/ivacaftor; lung and digestive microbiota and inflammation
MeSH Terms: conditions — Cystic Fibrosis; Inflammation | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with cystic fibrosis (Experimental): patients with cystic fibrosis before and one year after the start of treatment with elexacaftor/tezacaftor/ivacaftor
  Interventions: Procedure: Sample collection

INTERVENTIONS:
Procedure: Sample collection — collection of sputum, stool and blood samples at baseline, 6 months and 1 year after baseline

SUMMARY:
Cystic fibrosis is a systemic disease, which affects in particular the respiratory and digestive systems of patients, sites of chronic inflammation.

A new combination of elexacaftor/tezacaftor/ivacaftor has proven its efficacy for the treatment of patients aged 12 years and over with two F508del mutations or a so-called "minimal function" mutation associated with one F508del mutation. European marketing authorization was obtained in August 2020 and access in France should therefore arrive soon. Given that this treatment targets new mutations and that the efficacy seems greater than with LUM/IVA, it is important to assess its impact on the microbiota and the pulmonary and digestive inflammation of patients.

It is therefore a question of taking advantage of the experience of the Lum-Iva-Biota cohort, and the validated and operational sample circuit established in the various participating centers to set up a biological collection for the collection and storage of sputum and stools of patients during the first year of treatment with elexacaftor/tezacaftor/ivacaftor, in order to study the effect of treatment on the lung and digestive microbiota/mycobiota and inflammation.

DETAILED DESCRIPTION:
Cystic fibrosis is a systemic disease, which affects in particular the respiratory and digestive systems of patients, sites of chronic inflammation. It has also been shown that in these patients, the pulmonary and intestinal microbiota were distinct from those of healthy subjects and that the progression of the disease was associated with alterations in these microbiota. In addition, numerous data suggest the existence of an "intestinal-lung axis" and therefore encourage studying these two organs in parallel and not separately.

The management of cystic fibrosis has been marked in recent years by the appearance of CFTR modulators, in particular the combination lumacaftor/ivacaftor (LUM/IVA) (for patients homozygous F508del). The criteria for evaluating the efficacy of these treatments are based on the change in FEV (forced expiratory volume in 1 second), the number of exacerbations, body mass index or quality of life. However, it is essential to be able to document the effect of these treatments on the lung and digestive microbiota and inflammation. Since 2016, we have set up the national "Lum-Iva-Biota" cohort and have been able to show that the effect of LUM/IVA on the pulmonary microbiota was more marked in patients not previously colonized with P. aeruginosa.

A new combination of elexacaftor/tezacaftor/ivacaftor has proven its efficacy for the treatment of patients aged 12 years and over with two F508del mutations or a so-called "minimal function" mutation associated with one F508del mutation. European marketing authorization was obtained in August 2020 and access in France should therefore arrive soon. Given that this treatment targets new mutations and that the efficacy seems greater than with LUM/IVA, it is important to assess its impact on the microbiota and the pulmonary and digestive inflammation of patients.

It is therefore a question of taking advantage of the experience of the Lum-Iva-Biota cohort, and the validated and operational sample circuit established in the various participating centers to set up a biological collection for the collection and storage of sputum and stools of patients during the first year of treatment with elexacaftor/tezacaftor/ivacaftor, in order to study the effect of treatment on the lung and digestive microbiota/mycobiota and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* To have cystic fibrosis (sweat test > 60 mmol/l);
* Carrier of at least one DeltaF508 mutation;
* Be followed in the current care by a participant in the CRCM study;
* Start treatment with elexacaftor/tezacaftor/ivacaftor in routine care, according to the indications in the Marketing Authorization at the time of inclusion;
* Be of the age specified in the marketing authorization in force;
* Person affiliated or beneficiary of a social security scheme;
* Consent obtained by the patient (for adult patients) or the holders of parental authority (for minor patients) before any examination required by the research and oral and/or written consent by the participant (depending on his or her age) .
* Patient agreeing to take part in cohort follow-up studies of patients treated with elexacaftor/tezacaftor/ivacaftor, included in the French cystic fibrosis register (cf. Study by Pr BURGEL and/or MODUL CF).

Exclusion Criteria:

* Start of treatment with elexacaftor/tezacaftor/ivacaftor as part of a therapeutic trial.
* Patient already on CFTR modulator (including lumacaftor/ivacaftor)
* Vulnerable people (pregnant woman, person under guardianship/curators)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 253 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-09-13 (Estimated); Study Completion 2024-09-13 (Estimated)

PRIMARY OUTCOMES:
composition of the digestive bacterial microbiota | 12 months after baseline (treatment initiation)
  composition of the digestive, bacterial microbiota, at 12 months of treatment

SECONDARY OUTCOMES:
composition of the pulmonary bacterial microbiota | 12 months after baseline (treatment initiation)
  composition of the pulmonary bacterialmicrobiota, at 12 months of treatment
composition of the pulmonary bacterial microbiota | at baseline (treatment initiation)
  composition of the pulmonary bacterialmicrobiota at baseline
composition of the digestive fungal microbiota | 12 months after baseline (treatment initiation)
  composition of the digestive fungal microbiota, at 12 months of treatment
composition of the digestive fungal microbiota | at baseline (treatment initiation)
  composition of the digestive fungal microbiota at baseline
composition of the pulmonary fungal microbiota | 12 months after baseline (treatment initiation)
  composition of the pulmonary fungal microbiota, at 12 months of treatment
composition of the pulmonary fungal microbiota | at baseline (treatment initiation)
  composition of the pulmonary fungal microbiota at baseline
composition of the digestive, bacterial microbiota | at baseline (treatment initiation)
  composition of the digestive, bacterial microbiota at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Enaud, MDPhD, Principal Investigator — University Hospital, Bordeaux
Locations (15):
- France (15):
  - CHU de Bordeaux - CRCM pédiatrique, Bordeaux
  - CHU de Grenoble Alpes CRCM pédiatrique, Grenoble
  - CHRU de Lille CRCM Pédiatrique, Lille
  - CHU de Limoges CRCM Limousin, Limoges
  - Hospices Civils de Lyon Service de pédiatrie, allergologie et mucoviscidose, Lyon
  - AP-HM CRCM pédiatrique, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nice, Nice
  - AP-HP CRCM Robert debré, Paris
  - AP-PH Hopital Cochin service de pédiatrie, Paris
  - APHP Hopital Necker, Paris
  - Fondation Ildys, Roscoff Centre Hélio Marin - Clinique "Mucoviscidose", Roscoff
  - CHU de Rouen, Rouen
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No